CLINICAL TRIAL: NCT01178983
Title: Efficacy of Telerehabilitation Intervention Program Using Telebiofeedback Among Computer Operators
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Merav Golombowicz, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-10-7334-RP-CTIL
Record Dates: First submitted 2010-08-09; First posted 2010-08-10 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Work Related Musculoskeletal Disorders
Keywords: work related musculoskeletal disorders (WRMSD) among computer operators
MeSH Terms: interventions — Electromyography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- telebiofeedback (Experimental)
  Interventions: Device: surface electromyography
- biofeedback (Active Comparator)
  Interventions: Device: surface electromyography

INTERVENTIONS:
Device: surface electromyography — Surface electromyography (SEMG) telebiofeedback
  Arms: telebiofeedback
Device: surface electromyography — conventional biofeedback
  Arms: biofeedback

SUMMARY:
In the recent decades, with technology development, computer workstation has become fundamental both at work and at home environments, and is now used routinely for many purposes. Musculoskeletal disorders (MSD) are most often characterized by backaches, neck and upper extremities pain, discomfort and pain in joints, muscles and soft tissues. Since it has been found that many musculoskeletal disorders are connected, among others, to biomechanical and psychosocial factors relating to a person's work environment, the literature refers to them as Work Related MSD (WRMSD). Risk factors correlated with WRMSD include repetitive motions, awkward positions or static muscle loading over prolonged periods of time, use of high keystroke force, direct mechanical pressure, vibration and extreme temperatures. Computer operators found to be sitting statically for a long time in front of the computer and keyboard, with limited options of changing body position. Psychosocial factors have also been implicated in the workstation musculoskeletal disorders with computer operators. Workers with WRMSD may suffer from persistent pain, loss of function and work disability. Therefore, it may include changes in the employment and earnings for injured workers. The complex nature of these injuries suggests that workplace rehabilitation interventions are a crucial aspect of treatment management.

The main objective of this study is to explore the use of biofeedback intervention, based on tele-rehabilitation principle, with computer operators suffer from WRMSD. Treatment efficacy will be tested by use of RULA (Rapid Upper Limb Assessment) method. Data analysis will be done by ANOVA Repeated Measures.

Hypothesis: Biofeedback intervention, based on tele-rehabilitation principle, will be found effective with computer operators suffer from WRMSD.

ELIGIBILITY:
Inclusion Criteria:

* computer operators who spend more than 4 hours a day working with computer
* computer operators who suffer from pain and inconvenience or injury in upper limbs, such as Lateral Epicondylitis, de Quervain disease, Carpal Tunnel Syndrome (CTS), Ulnar Tunnel Syndrome, Flexor-Extensor peritendinitis or teno-synovitis of the forearm-wrist region.

Exclusion Criteria:

* subjects who suffer from neurological injuries
* subjects who suffer from orthopedic injuries or other metabolic or autoimmune diseases, that cause joint oedema or hand numbness (pregnancy, diabetes, heart disease and arthritis).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Posture at work environment measured by Rapid Upper LImb Assessment (RULA) | 15 months

SECONDARY OUTCOMES:
Musculoskeletal Disorders (MSD) - pain and inconvenience | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Merav Golombowicz, BOT, Study Chair — Upper Limb Rehabilitation Center
Locations (1):
- Sheba Tel Hashomer hospital - upper limb rehabilitation center, Ramat Gan, Ramat Gan, Israel